CLINICAL TRIAL: NCT01893398
Title: Multistimulation Group Therapy in Mild to Moderate Alzheimer's Disease
Brief Title: Multistimulation Group Therapy for Alzheimer's Disease
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Fondazione Don Carlo Gnocchi Onlus (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single
Other Study IDs: FdG_AD_01
Record Dates: First submitted 2013-06-24; First posted 2013-07-09 (Estimated); Last update posted 2013-07-09 (Estimated); Status verified 2013-06

CONDITIONS: Alzheimer's Disease
MeSH Terms: conditions — Alzheimer Disease

STUDY DESIGN:
Who Masked: Outcomes Assessor

ARMS (2):
- rehabilitation (MST) program (Experimental): The Multidimensional Stimulation group therapy (MST) involved three levels of treatment. The first level was focused on PWA, the second level involved the caregiver, while the third one the dyad PWA-caregiver.
  Interventions: Other: Multidimensional stimulation group therapy
- Usual care program (No Intervention): Usual care PWA program

INTERVENTIONS:
Other: Multidimensional stimulation group therapy — The MST program involved three levels of treatment. The first level was focused on PWA, the second level involved the caregiver, while the third one the dyad PWA-caregiver.
  Arms: rehabilitation (MST) program

SUMMARY:
Our previous findings support the notion that group activity program, based on cognitive stimulation, recreational-occupational activities and physical-psychomotor exercises, can lead to an improvement in behavioral aspects for people with Alzheimer's Disease (AD).

The purpose of this study is to clarify the efficacy of a rehabilitation program in outpatients affected by AD in mild to moderate stages.

ELIGIBILITY:
Inclusion Criteria:

* diagnosis of possible/probable AD
* mild to moderate stage of AD (MMSE score of 15 - 24)and CDR score of 1-2
* range years in age (65-85) and in school attendance (5-17)
* right handed

Exclusion Criteria:

* severe aphasia (Token test score < 20)
* severe auditory and/or visual loss
* overt severe behavioral disturbances (delusions, hallucinations, agitation)
* recent (three month before the MST) introduction or dose modification of the following pharmacological treatments: cholinesterase inhibitor, memantine, antidepressant or antipsychotic drugs.

Ages: 65 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Enrollment: 60 (Actual)
Dates: Start 2010-01; Primary Completion 2012-12 (Actual)

PRIMARY OUTCOMES:
Change from baseline in behavioral level | Baseline, 10ws, 22ws
  Neuropsychiatric Inventory scale
Change from baseline in cognitive level | Baseline, 10ws, 22 ws
  ADAS cog scale
Change from baseline in quality of life | baseline, 10ws,22 ws
  SF36 questionaire

OTHER OUTCOMES:
Functional MRI | baseline, 10 ws
  Change from baseline in brain functioning. We used fMRI with cognitive task to detect possible changes (10 ws versus baseline) in brain activation patterns in PWA as a surrogate biomarker of efficacy.

CONTACTS AND LOCATIONS:
Locations (1):
- IRCCS, S Maria Nascente, FOndazione don Gnocchi, Milan, Italy

REFERENCES:
- [Background] Farina E, Mantovani F, Fioravanti R, Pignatti R, Chiavari L, Imbornone E, Olivotto F, Alberoni M, Mariani C, Nemni R. Evaluating two group programmes of cognitive training in mild-to-moderate AD: is there any difference between a 'global' stimulation and a 'cognitive-specific' one? Aging Ment Health. 2006 May;10(3):211-8. doi: 10.1080/13607860500409492. PMID 16777648
- [Background] Farina E, Fioravanti R, Chiavari L, Imbornone E, Alberoni M, Pomati S, Pinardi G, Pignatti R, Mariani C. Comparing two programs of cognitive training in Alzheimer's disease: a pilot study. Acta Neurol Scand. 2002 May;105(5):365-71. doi: 10.1034/j.1600-0404.2002.01086.x. PMID 11982487
- See also: Related Info — http://www.dongnocchi.it/